CLINICAL TRIAL: NCT02543242
Title: Effectiveness of the Intone Pelvic Floor Device for Urinary Incontinence
Brief Title: InTone for Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: InTone
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence; Stress Urinary Incontinence; Urge Incontinence; Mixed Urinary Incontience; Female Pelvic Health
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress; Urinary Incontinence, Urge | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Participants will undergo the InTone TM (InControl Medical, LLC) medical device treatment for Urinary Incontinence. The frequency of treatment is once/day (12 minutes), 5-6 days/week. The route of administration is vaginal.
  Interventions: Device: InToneTM (InControl Medical, LLC) - Medical Device

INTERVENTIONS:
Device: InToneTM (InControl Medical, LLC) - Medical Device

SUMMARY:
The rationale for the conduct of this study is that the Intone device (along with pelvic physiotherapy) can be used to help females suffering from urinary stress incontinence by using electrical stimulation and biofeedback during pelvic floor muscle training. This investigation is important because it can aid in the greater acceptance and development of non-surgical treatments for Stress Urinary Incontinence if these areas are looked into. The study results will address if the Intone device is beneficial and promotes long-term improvement in women that suffer from urinary incontinence.

DETAILED DESCRIPTION:
Urinary incontinence is very common in women and is linked to a reduced quality of life (Corcos et al., 2002). The three main types of urinary incontinence are Stress Urinary Incontinence (SUI), Urge Urinary Incontinence (UUI) and Mixed Urinary Incontinence (MUI). SUI and UUI involve losing urine involuntarily. In SUI this is during either effortful motion such as coughing or sneezing, or in UUI is associated with a feeling of urgency. Urinary incontinence has various treatment options including: surgery, medication, pelvic floor muscle exercises and electrical stimulation (Norton & Brubaker, 2006).

The most common physiotherapy treatment used for women with urinary incontinence is pelvic floor muscle training (Dumoulin & Hay-Smith, 2010). Several studies have investigated the effects of PFMT in comparison to other treatments such as no treatment and vaginal cones. They found that women in the PFMT group reported more improvement and better quality of life than women in other treatment groups. The PFMT group also had fewer daily incontinence episodes and less leakage (Bø, Talseth, & Holme, 1999; Dumoulin & Hay-Smith, 2010).

Electrical stimulation of the pelvic floor muscles is another treatment for urinary incontinence, and may often be combined with PFMT. Success rates of electrical stimulation in treating urinary incontinence range from 50-90% (Bent et al., 1993; Erikson, Bergmann, & Mjølnerød, 1987; Fall, 1984; Pelvnik et al., 1986).

A new product has been developed called InTone which combines PFMT, electrical stimulation and biofeedback. This device is inserted into the vagina and facilitates PFMT while providing electrical stimulation and biofeedback to the patient. This study will examine the effectiveness of the InTone device in treating urinary incontinence in women.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Between ages 18-70
* Diagnosed with Stress Urinary Incontinence (SUI), Urge Urinary Incontinence (UUI), or Mixed Urinary Incontinence (MUI)

Exclusion Criteria:

* Incontinence of less than 6 months
* pregnancy or delivery within 6 weeks
* vaginal or pelvic surgery within previous 6 months
* pelvic organ prolapse greater than stage 2 (based on POP-Q)
* active UTI or history of recurrent UTIs (more than 3 in a year)
* recurrent vaginitis (bacterial/fungal)
* pelvic pain/painful bladder syndrome
* implanted cardiac device or untreated cardiac arrhythmi
* Underlying neurologic/neuromuscular disorder, or inadequate vaginal caliber (can't accommodate device).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Pad Test Weighting | up to 26 weeks
  urine voiding measure

SECONDARY OUTCOMES:
Urinary Distress Inventory (UDI-6) | screening, Device Set up/Training Day, 2, 6, 14, 26 weeks from set up.
  Questionnaire that assesses symptom distress and the impact on daily life of urinary incontinence
Incontinence Impact Questionnaire Short Form (IIQ-7) | screening, Device Set up/Training Day, 2, 6, 14, 26 weeks from set up.
  Assesses symptom distress and the impact on daily life of urinary incontinence
Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) | screening, Device Set up/Training Day, 2, 6, 14, 26 weeks from set up.
  Evaluates sexual function in women with pelvic organ prolapse and/or urinary incontinence.
Urinary Incontinence Quality of Life Scale (IQOL) | screening, Device Set up/Training Day, 2, 6, 14, 26 weeks from set up.
  A self-reported quality of life measure specific to urinary incontinence (UI),
International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ UI SF) | screening, Device Set up/Training Day, 2, 6, 14, 26 weeks from set up.
  A subjective measure of severity of urinary loss and quality of life for those with urinary incontinence.
48 Hour Bladder Diary | up to 6 months follow-up
  A diary containing details of every void. The time, amount leaked and activity during the leakage are recorded for 48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Dean S Elterman, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network (Altum Health), Toronto, Ontario, Canada

REFERENCES:
- [Background] Brubaker L, Benson JT, Bent A, Clark A, Shott S. Transvaginal electrical stimulation for female urinary incontinence. Am J Obstet Gynecol. 1997 Sep;177(3):536-40. doi: 10.1016/s0002-9378(97)70142-x. PMID 9322620
- [Background] Corcos J, Beaulieu S, Donovan J, Naughton M, Gotoh M; Symptom Quality of Life Assesment Committee of the First International Consultation on Incontinence. Quality of life assessment in men and women with urinary incontinence. J Urol. 2002 Sep;168(3):896-905. doi: 10.1016/S0022-5347(05)64540-5. PMID 12187188
- [Background] Dumoulin C, Hay-Smith J, Habee-Seguin GM, Mercier J. Pelvic floor muscle training versus no treatment, or inactive control treatments, for urinary incontinence in women: a short version Cochrane systematic review with meta-analysis. Neurourol Urodyn. 2015 Apr;34(4):300-8. doi: 10.1002/nau.22700. Epub 2014 Nov 18. PMID 25408383
- [Background] Eriksen BC, Bergmann S, Mjolnerod OK. Effect of anal electrostimulation with the 'Incontan' device in women with urinary incontinence. Br J Obstet Gynaecol. 1987 Feb;94(2):147-56. doi: 10.1111/j.1471-0528.1987.tb02342.x. PMID 3493802
- [Background] Fall M. Does electrostimulation cure urinary incontinence? J Urol. 1984 Apr;131(4):664-7. doi: 10.1016/s0022-5347(17)50566-2. PMID 6608590
- [Background] Bo K, Talseth T, Holme I. Single blind, randomised controlled trial of pelvic floor exercises, electrical stimulation, vaginal cones, and no treatment in management of genuine stress incontinence in women. BMJ. 1999 Feb 20;318(7182):487-93. doi: 10.1136/bmj.318.7182.487. PMID 10024253
- [Background] Norton P, Brubaker L. Urinary incontinence in women. Lancet. 2006 Jan 7;367(9504):57-67. doi: 10.1016/S0140-6736(06)67925-7. PMID 16399154
- [Background] Tjelum KB, Lose G, Abel I, Pedersen LM. [Electrostimulation of the pelvic floor muscles in urinary incontinence]. Ugeskr Laeger. 1994 Apr 11;156(15):2214-6. Danish. PMID 8016945